CLINICAL TRIAL: NCT04857996
Title: A Phase 2a, Prospective, Multicenter, Randomized, Double Masked, Sham-Controlled Study to Assess the Safety, Tolerability and Evidence of Activity of a Single Intravitreal Injection of UBX1325 in Patients With Diabetic Macular Edema
Brief Title: Safety, Tolerability and Evidence of Activity Study of UBX1325 in Patients With Diabetic Macular Edema (BEHOLD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Unity Biotechnology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UBX1325-02
Record Dates: First submitted 2021-04-21; First posted 2021-04-23 (Actual); Results first posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-04

CONDITIONS: Diabetic Macular Edema (DME)
Keywords: Retinal disease; Macular edema; Diabetes mellitus; Diabetic macular edema
MeSH Terms: conditions — Retinal Diseases; Macular Edema; Diabetes Mellitus | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: This study will be double masked, so patients and Investigators are masked to the treatment assigned, while certain roles at the site and at the Sponsor are unmasked. Sites will have a qualified injector who is unmasked to perform the study treatment injection or sham procedure, as well as certain post-injection assessments on Day 1 only.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- UBX1325 (Experimental)
  Interventions: Drug: UBX1325
- Sham Control (Sham Comparator)
  Interventions: Other: Sham

INTERVENTIONS:
Drug: UBX1325 — Patients will be administered a single 50 μL UBX1325 IVT injection
  Arms: UBX1325
Other: Sham — Sham procedure
  Arms: Sham Control

SUMMARY:
This study is intended to assess the exposure, safety, biological activity, and durability of UBX1325, a phosphate pro-drug, and its active parent molecule (UBX0601) following a single intravitreal (IVT) injection of UBX1325 in patients with diabetic macular edema (DME).

DETAILED DESCRIPTION:
This is a Phase 2a Proof-of-Concept (POC) study. The study will enroll approximately 62 patients randomized 1:1 into either the UBX1325 or sham study arms, in order to assess safety and tolerability as well as impact on visual function and retinal anatomy. Patients will be followed for 24 weeks for the primary outcome measure and for an additional 24 weeks (48 weeks total) for the secondary outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 18 years.
* Diabetic retinopathy patients (nonproliferative (NPDR) and proliferative (PDR)) with DME (ETDRS-DRSS Score at 65C [or DR severity level of 8]or less severe as determined by a Central Reading Center), who had at least 2 anti-VEGF intravitreal (IVT) injections (one or more of the following agents: aflibercept, bevacizumab or ranibizumab) in the preceding 6 months prior to Day 1, with the last anti-VEGF given between 3 and 6 weeks prior to Day 1.
* Center-involved DME with central subfield thickness (CST) ≥300 µm on SD-OCT at Screening
* BCVA in the study eye (most affected) of 73 to 20 ETDRS letters (equivalent to 20/40 to 20/400 on the Snellen chart) at Screening and at Day 1.

Exclusion Criteria:

* Concurrent disease in the study eye or structural damage, other than DME, that could compromise BCVA, prevent BCVA improvement, require medical or surgical intervention during the study period, confound interpretation of the results, or interfere with assessment of toxicity or color fundus photography (CFP) in the study eye.
* Any ocular/intraocular/periocular infection or inflammation in either eye in the past 4 weeks prior to screening
* History of vitreous hemorrhage in the study eye within 2 months prior to Screening
* Any condition, including laboratory findings and findings in the medical history or in the pre-study assessments, that, in the opinion of the Investigator, constitutes a risk or contraindication for participation in the study or that could interfere with the study objectives, conduct, or evaluation or prevent the patient from fully participating in all aspects of the study
* Significant media opacities, including cataract, which might interfere with VA, assessment of toxicity, or fundus imaging

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2021-06-25 (Actual); Primary Completion 2023-04-06 (Actual); Study Completion 2023-04-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Klier, MD, MPH, Study Director — Unity Biotechnology, Inc.
Locations (22):
- United States (19):
  - Retinal Research Institute, LLC, Phoenix, Arizona
  - California Retina Consultants, Bakersfield, California
  - The Retina Partners, Encino, California
  - Salehi Retina Institute Inc., Huntington Beach, California
  - Loma Linda University, Loma Linda, California
  - California Retina Consultants, Oxnard, California
  - Advanced Vision Research Institute, Longmont, Colorado
  - Bascom Palmer Eye Institute, Miami, Florida
  - MedEye Associates, Miami, Florida
  - Northwestern Medical Group, Chicago, Illinois
  - MidWest Eye Institute, Indianapolis, Indiana
  - Cumberland Valley Retina Consultants, Hagerstown, Maryland
  - Mass Eye and Ear Institute, Boston, Massachusetts
  - Sierra Eye Associates, Reno, Nevada
  - New York Eye and Ear Infirmary, New York, New York
  - EyeHealth Northwest, Portland, Oregon
  - Retina Consultants of Carolina, PA, Greenville, South Carolina
  - Valley Retina Institute, P.A., McAllen, Texas
  - Retina Center of Texas, Southlake, Texas
- Canada (3):
  - Alberta Retina Research Corporation, Edmonton, Alberta
  - Toronto Retina Institute, North York, Ontario
  - Hopital Maisonneuve-Rosemont, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Klier S, Dananberg J, Masaki L, Bhisitkul RB, Khanani AM, Maturi R, Salehi-Had H, Mallinckrodt CH, Rathmell JM, Ghosh A, Sapieha P. Safety and Efficacy of Senolytic UBX1325 in Diabetic Macular Edema. NEJM Evid. 2025 May;4(5):EVIDoa2400009. doi: 10.1056/EVIDoa2400009. Epub 2025 Apr 22. PMID 40261111

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: each participant contributed only one study eye
Units Other Than Participants: study eye
Groups:
- UBX1325: UBX1325: Patients will be administered a single 10 μg UBX1325 IVT injection
Period: Overall Study
Arm/Group | Sham Control | UBX1325
Started | 33; 33 study eye | 32; 32 study eye
Completed | 26; 26 study eye | 24; 24 study eye
Not Completed | 7; 7 study eye | 8; 8 study eye
Not completed — Completed 24 weeks before study extension to 48 weeks was available as per Protocol version 4.0 | 4 | 5
Not completed — Lost to Follow-up | 1 | 3
Not completed — Site Closure | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sham Control | UBX1325 | Total
Number analyzed (Participants) | 33 | 32 | 65
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.4 (9.09) | 63.6 (9.33) | 62.5 (9.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 8 | 21
  Male | 20 | 24 | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 8 | 12
  Not Hispanic or Latino | 29 | 24 | 53
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 3 | 1 | 4
  Black or African American | 3 | 2 | 5
  White | 25 | 24 | 49
  Other | 2 | 3 | 5
  Not reported | 0 | 1 | 1
Study Eye [Count of Participants; unit: Participants]
  Left Eye | 11 | 18 | 29
  Right eye | 22 | 14 | 36
Eye Color [Count of Participants; unit: Participants]
  Blue | 8 | 10 | 18
  Brown | 18 | 19 | 37
  Green | 0 | 2 | 2
  Hazel | 7 | 0 | 7
  Other | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Systemic Safety and Tolerability of a Single IVT Injection of UBX1325.
Description: The systemic safety and tolerability is evaluated by incidence of Treatment Emergent Adverse Events (TEAEs) by System organ class Preferred Term.
Time Frame: 48 weeks
Population: The Safety Analysis Set includes all patients who received a single IVT treatment of UBX1325 or sham. Summary statistics are frequency (percentage of column total).
Measure: Count of Participants; unit: Participants
Groups:
- Overall: Overall participants that received either Sham or UBX1325 10μg treatment
Arm/Group | Sham Control | UBX1325 | Overall
Number analyzed (Participants) | 33 | 32 | 65
Participants
  Subjects with at Least One Serious TEAE | 4 | 5 | 9
  Blood and lymphatic system disorders - Anemia | 0 | 1 | 1
  Cardiac disorders - Atrial fibrillation | 0 | 1 | 1
  Cardiac disorders - Coronary artery occlusion | 0 | 1 | 1
  Eye disorders-Visual acuity reduced | 1 | 0 | 1
  Eye disorders - Vitreous haemorrhage | 1 | 0 | 1
  Infections and infestations - Cellulitis | 0 | 1 | 1
  Infections and infestations - Pneumonia | 0 | 1 | 1
  Injury, poisoning and procedural complication - Ankle fracture | 0 | 1 | 1
  Injury, poisoning and procedural complication- Skin abrasion | 0 | 1 | 1
  Nervous system disorders - Cerebrovascular accident | 1 | 0 | 1
  Vascular disorders - Aortic stenosis | 1 | 0 | 1

2. Primary Outcome: Ocular Safety and Tolerability of a Single IVT Injection of UBX1325
Description: Ocular Safety is evaluated by incidence of Treatment Emergent Adverse Events (TEAEs).
  Ocular TEAEs consisted of progression of disease or were related to the IVT injection component of the UBX1325 drug administration process
Time Frame: Up to Week 12, 24 and 48 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Overall: Overall participants that received either Sham or UBX132510μg treatment
Arm/Group | Sham Control | UBX1325 | Overall
Number analyzed (Participants) | 33 | 32 | 65
Participants
  Subjects with At Least One Ocular TEAE in Study Eye | 28 | 23 | 51
  Eye disorders | 28 | 23 | 51
  Diabetic retinal oedema | 18 | 14 | 32
  Conjunctival haemorrhage | 2 | 8 | 10
  Vitreous haemorrhage | 5 | 2 | 7
  Macular thickening | 2 | 1 | 3
  Retinal oedema | 2 | 1 | 3
  Cataract subcapsular | 1 | 1 | 2
  Eye irritation | 0 | 2 | 2
  Cataract nuclear | 1 | 1 | 2
  Visual acuity reduced | 2 | 0 | 2
  Anterior chamber pigmentation | 0 | 1 | 1
  Conjunctival hyperaemia | 1 | 0 | 1
  Dry eye | 0 | 1 | 1
  Foreign body sensation in eyes | 1 | 0 | 0
  Meibomian gland dysfunction | 0 | 1 | 1
  Ocular hypertension | 0 | 1 | 1
  Posterior capsule opacification | 1 | 0 | 1
  Punctate keratitis | 0 | 1 | 1
  Retinal exudates | 1 | 0 | 1
  Retinal haemorrhage | 0 | 1 | 1
  Vitreous floaters | 1 | 0 | 1

3. Secondary Outcome: Changes in Best Corrected Visual Acuity (BCVA) From Baseline
Description: Best Corrected Visual Acuity was assessed using the ETDRS chart starting at 4 meters
Time Frame: Week 12, 24 and 48
Population: MMRM Model for BCVA Change from Baseline (Hypothetical Strategy) Full Analysis Set. The hypothetical strategy included all subjects but excluded observations post-rescue.
  The Full Analysis Set includes all randomized subjects who received a single IVT treatment of UBX1325 or sham, have a baseline BCVA assessment, and at least one post-baseline BCVA assessment.
Measure: Least Squares Mean (Standard Error); unit: ETDRS Letters
Arm/Group | Sham Control | UBX1325
Number analyzed (Participants) | 32 | 32
ETDRS Letters
  Week 12: number analyzed (Participants) | 21 | 24
  Week 12 | 1.5 (1.68) | 4.7 (1.59)
  Week 24: number analyzed (Participants) | 14 | 16
  Week 24 | -1.4 (1.99) | 6.7 (1.88)
  Week 48: number analyzed (Participants) | 6 | 12
  Week 48 | 0.6 (2.90) | 6.2 (2.12)

ADVERSE EVENTS:
Time Frame: up to 48 weeks
Arm/Group | Sham Control | UBX1325
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/32
Serious Adverse Events (participants affected / at risk) | 4/33 | 5/32
Other Adverse Events (participants affected / at risk) | 31/33 | 24/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sham Control (N=33) | UBX1325 (N=32)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery occlusion (Cardiac disorders) | 0 (0) | 1 (1)
Visual acuity reduced (Eye disorders) | 1 (1) | 0 (0)
Vitreous haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Aortic stenosis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sham Control (N=33) | UBX1325 (N=32)
Diabetic retinal oedema (Eye disorders) | 19 (19) | 17 (17)
Conjunctival haemorrhage (Eye disorders) | 2 (2) | 8 (8)
Cataract subcapsular (Eye disorders) | 2 (2) | 1 (1)
Vitreous haemorrhage (Eye disorders) | 4 (4) | 3 (3)
Eye irritation (Eye disorders) | 0 (0) | 2 (2)
Macular thickening (Eye disorders) | 2 (2) | 1 (1)
Posterior capsule opacification (Eye disorders) | 3 (3) | 0 (0)
Retinal oedema (Eye disorders) | 2 (2) | 1 (1)
Visual acuity reduced (Eye disorders) | 2 (2) | 0 (0)
COVID-19 (Infections and infestations) | 5 (5) | 4 (4)
Nasopharyngitis (Infections and infestations) | 3 (3) | 1 (1)
Electrocardiogram abnormal (Investigations) | 0 (0) | 2 (2)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 1 (1)
Depression (Psychiatric disorders) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 3 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-02-14): https://cdn.clinicaltrials.gov/large-docs/96/NCT04857996/Prot_002.pdf
  • Statistical Analysis Plan (2022-07-22): https://cdn.clinicaltrials.gov/large-docs/96/NCT04857996/SAP_003.pdf